CLINICAL TRIAL: NCT00222937
Title: Efficacy of Voice Therapy for Phonotrauma in Teachers
Brief Title: Voice Therapy for Teachers With Voice Problems
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Kittie Verdolini Abbott, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: #0304044
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2016-01

CONDITIONS: Phonotrauma
Keywords: Voice Problems; Voice Disorders
MeSH Terms: conditions — Voice Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Patients are enrolled in Lessac-Madsen Resonant Voice Therapy.
  Interventions: Behavioral: Lessac-Madsen Resonant Voice Therapy
- B (Experimental): Patients are enrolled in Casper Based Confidential Flow Therapy.
  Interventions: Behavioral: Casper-Based Confidential Flow Therapy

INTERVENTIONS:
Behavioral: Lessac-Madsen Resonant Voice Therapy — Patients receive 8 sessions of therapy over a course of 4 weeks, with one double session per week.
  Arms: A
Behavioral: Casper-Based Confidential Flow Therapy — Patients receive 8 sessions of therapy over a course of 4 weeks, with one double session per week.
  Arms: B

SUMMARY:
The study compares two different forms of voice therapy, Lessac-Madsen Resonant Voice Therapy and Casper-Based Confidential Flow Therapy. The target population are teachers because they have the highest risk for developing voice problems. For this study the investigators are primarily interested in seeing if Lessac-Madsen Resonant Voice Therapy (LMRVT) and Casper-Based Confidential Flow Therapy (CBCFT) are equally effective at improving vocal functioning in teachers with phonotrauma, as assessed by the Voice Handicap Index (VHI).

ELIGIBILITY:
Inclusion Criteria:

* Full or part time teacher including college professor, daycare and preschool
* 21 years of age and older
* Complaints of voice problems declared to be lasting continuously for one month or more
* Any structural or functional change to the larynx that appears related to phonation,including bilateral or unilateral lesions (assuming normal overlying epithelium based on clinical examination), non-specific edema, or erythema that appear by clinical history related to phonation, or primary muscle tension dysphonia or other condition related to phonation without lesions
* No concurrent ear, nose and/or throat diagnoses, e.g. acute allergies, except for chronic allergies, sinusitis, and laryngopharyngeal reflux disease (LPR)
* No vocal fold hemorrhage
* No known degenerative medical conditions (e.g., degenerative neuromuscular disease, malignant process undergoing treatment or with less than 5 years remission, uncontrolled systemic disease (e.g., auto immune disease, or hormonal condition)
* Normal hearing to 30 dB at 1000Hz - 3000Hz in the better ear
* The participant is able to start therapy within 6 weeks of the initial evaluation and can be scheduled for 8 sessions (two per visit) in a 6-week time period
* Agreement by the participant to provide information regarding days missed from work during the previous year and the year following treatment

Exclusion Criteria:

* Known degenerative medical condition
* Concurrent ear-nose-throat diagnosis, e.g., acute allergies (but chronic allergies, sinusitis, and laryngopharyngeal reflux disease (LPR) are not exclusion criteria) and vocal fold hemorrhage
* Degenerative medical conditions that would exclude a participant from participation include, but are not limited to: degenerative neuromuscular disease, malignant process undergoing treatment or with less than 5 years remission, uncontrolled systemic disease (e.g. auto immune disease), or hormonal condition.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2005-10; Primary Completion 2009-06 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Score on Voice Handicap Index (VHI) | one year

SECONDARY OUTCOMES:
Does LMRVT contribute to the actual acquisition of "resonant voice" in speech? | one year
Do LMRVT or CBCFT improve laryngeal appearance? | one year
Do LMRVT or CBCFT improve conversational voice quality? | one year
Do LMRVT or CBCFT reduce the occurrence of laryngeal microsurgery? | one year
Do LMRVT or CBCFT reduce the number of workdays lost annually? | one year

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Verdolini, Ph.D., Principal Investigator — University of Pittsburgh; Clark Rosen, M.D., Study Director — University of Pittsburgh; Jackie Gartner-Schmidt, Ph.D., Study Director — University of Pittsburgh; Franca Benedicty Barton, M.S., Study Director — The Emmes Company, LLC
Locations (2):
- United States (2):
  - Massachusetts Eye & Ear Infirmary, Voice and Speech Laboratory, Boston, Massachusetts
  - University of Pittsburgh Medical Center, Voice Center, Pittsburgh, Pennsylvania